CLINICAL TRIAL: NCT05921773
Title: Clinical Evaluation of Functional Near-infrared Spectroscopy for Anxiety Monitoring and Neurofeedback.
Brief Title: Functional Near-infrared Spectroscopy for Anxiety Monitoring and Neurofeedback.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202302110DINA
Record Dates: First submitted 2023-06-13; First posted 2023-06-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GAD Patients with Intervention (Experimental): The feedback group will get real neurofeedback about changes in anxiety-related cerebral hemodynamics. AI-fNIRS neurofeedback will be provided 3 times a week, for a total of 4 weeks.
  Interventions: Device: AI-fNIRS neurofeedback device
- GAD Patients with Sham Controls (Sham Comparator): The sham group will be shown playbacks of someone's real feedback sessions. Sham AI-fNIRS neurofeedback will be provided 3 times a week, for a total of 4 weeks.
  Interventions: Device: AI-fNIRS neurofeedback device with sham signals

INTERVENTIONS:
Device: AI-fNIRS neurofeedback device — The device, with AI-fNIRS signals serving as brain monitor to indicate the level of anxiety, provides mindfulness training through visual and auditory cues to help participants modulate their brain activity, and thus alleviates anxious states.
  Arms: GAD Patients with Intervention
Device: AI-fNIRS neurofeedback device with sham signals — The sham control consists of playbacks of someone else's real AI-fNIRS neurofeedback and will be provided 3 times a week, for a total of 4 weeks.
  Arms: GAD Patients with Sham Controls

SUMMARY:
The objective of this subproject is to validate the efficacy of the fNIRS real-time anxiety monitoring and neurofeedback system. In the first year, the cerebral hemodynamics measured by commercial fNIRS during resting state and cognitive tasks from 60 generalized anxiety disorder (GAD) patients and 30 healthy subjects will be processed and analyzed using AI algorithms. The novel anxiety fNIRS biomarker will be identified and correlated to clinical anxiety scales (such as HARS and STAI). In the second year, the validity and responsiveness of the AI-fNIRS biomarker will be validated. The accuracy of using AI-fNIRS biomarker to predict the diagnosis of GAD (according to DSM-5) and anxiety rating scales will be calculated from 60 GAD patients and 30 healthy subjects. In the third year, a neurofeedback method using AI-fNIRS biomarkers to guide digital cognitive behavior therapy (dCBT) through visual/audio cues will be developed. A pilot study with 12 GAD patients will be performed to test the feasibility of mindfulness training during AI-fNIRS neurofeedback. In the fourth year, a large scale RCT will be performed to validate the therapeutic efficacy of AI-fNIRS neurofeedback dCBT in 40 patients with GAD. The protocol of using real-time AI-fNIRS biomarkers as a neurofeedback to augment mindfulness training will be optimized according to previous year.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with generalized anxiety disorder (GAD) by psychiatrists based on DSM-V.
* Native Chinese speakers.
* Right-handers.
* Normal vision without or after correction.
* Normal hearing and verbal expression.
* Regular returns of medical or psychological intervention during participation.

Exclusion Criteria:

* Being diagnosed with other major neurological or mental disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral hemodynamics from functional near-infrared spectroscopy (fNIRS) | Baseline, 4-week intervention, and 2 months after 4-week intervention.
  fNIRS is an optical brain monitoring technique. It serves as an ideal tool to record brain activities based on hemodynamics during various cognitive or motor tasks. The regions of interest are bihemispheric prefrontal cortices.
Change in severity of physiological and psychological anxious symptoms as assessed by Hamilton Anxiety Rating Scale (HARS) | Baseline, 4-week intervention, and 2 months after 4-week intervention.
  Hamilton Anxiety Rating Scale (HARS) is a frequently-used scale in clinical psychiatric fields to assess the severity of anxious symptoms. Conducted by well-trained clinicians, HARS consists of 14 items and can be classified into 2 domains: physiological and psychological anxious symptoms. The minimum and maximum values are 0 and 56 respectively, with higher scores represent worse outcomes.
Change in temporary and long-term anxiety levels as assessed by State-Trait Anxiety Inventory (STAI) | Baseline, 4-week intervention, and 2 months after 4-week intervention.
  State-Trait Anxiety Inventory (STAI) is a self-report measure of subjective feelings of anxiety. It consists of 2 subscales: state and trait anxiety, with the former characteristic of temporary states of emotion and the latter dealing with the frequency of anxiety and other related emotion in general conditions. The minimum and maximum values of each subscale are 20 and 80 respectively. The higher the score, the higher the level of anxiety.
Change in anxiety level as reported in Visual Analog Scale (VAS) | Baseline, 4-week intervention, and 2 months after 4-week intervention.
  VAS is a self-report measure. Participants are required to draw a 10 cm line representing their anxiety spectrum, and mark their subjective feelings of anxiety level on it, with the highest on the right end.
Change in physiological anxious symptoms indicated by Heart Rate Variability (HRV) | Baseline, 4-week intervention, and 2 months after 4-week intervention.
  Measured with NeXus-10MKII (Mind Media, the USA), HRV serves as a physiological index of anxiety. Subjects with anxiety will show lower HRV than healthy individuals.

SECONDARY OUTCOMES:
Change in severity of depressive symptoms as assessed by Hamilton Depression Rating Scale (HAM-D) | Baseline, 4-week intervention, and 2 months after 4-week intervention.
  The HAM-D consists of 17 items reflecting depressive symptoms, with higher scores indicating more severe depressive symptoms for that particular item. The total score ranges from 0 to 52.
Change in performance on emotional dual N-back task | Baseline, 4-week intervention, and 2 months after 4-week intervention.
  Facial expressions and colored emotional words are simultaneously presented a screen. Participants are required to remember the location of the image and the color of the word, while trying to ignore the facial expression and the emotional meaning of the word.
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline, 4-week intervention, and 2 months after 4-week intervention.
  PSQI is a self-report measure of sleep quality. It consists of 9 items and is related to 7 dimensions of sleep. The higher the score is, the worse the quality of sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan